CLINICAL TRIAL: NCT04528628
Title: Optimization of Diagnosis and Treatment of Depression Based on Multidimensional Clinical Assessment Classification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: RenJi Hospital (Other); Shanghai 10th People's Hospital (Other); Huashan Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Nanjing Medical University (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHZD2020PDH
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Serotonin; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MDD with melancholic features (Experimental)
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: Treatment as Usual; Combination Product: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) Combined with Magnetic Stimulations
- MDD with atypical features (Experimental)
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: Treatment as Usual; Combination Product: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) Combined with Magnetic Stimulations
- MDD with anxious distress (Experimental)
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: Treatment as Usual; Combination Product: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) Combined with Magnetic Stimulations
- MDD (overall) (Experimental)
  Interventions: Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors); Drug: Treatment as Usual; Combination Product: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) Combined with Magnetic Stimulations

INTERVENTIONS:
Drug: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) — Patients will be treated with one kind of selective serotonin reuptake inhibitors/ serotonin and norepinephrine reuptake inhibitors. Dose is titrated to the minimum effective dose within 2 weeks. Benzodiazepines can be used for a short period lasting no more than 2 weeks.
Drug: Treatment as Usual — The research doctor discusses the treatment plan with the patient, and therapies and drugs are not limited.
Combination Product: SSRIs/SNRIs (Selective Serotonin Reuptake Inhibitors/ Serotonin and Norepinephrine Reuptake Inhibitors) Combined with Magnetic Stimulations — Drug therapies are the same as the SSRIs/SNRIs monotherapy group. Patients will randomly receive one kind of magnetic stimulations including repetitive transcranial magnetic stimulation (rTMS), continuous theta burst stimulation(cTBS) and intermittent theta burst stimulation (iTBS) at a ratio of 1:1:1.

SUMMARY:
Major depressive disorder (MDD) characterized by high prevalence, high recurrence rate and high disability rate is a mental illness with the heaviest burden and has become a major public health issue in China and the world. Great challenges in diagnosis and treatment of depression consist of the complicated pathogenesis, a lack of objective diagnostic criteria, unsatisfactory treatment outcomes and poor treatment compliance. The previous studies of our research team showed that depression is affected by multiple factors. We could explore important markers for the diagnosis, treatment and prediction of treatment efficacy in depressed patients' data collected from different dimensions including immunometabolism, brain electrophysiology, brain structure and functional neural circuits, neuropsychology and psychophysiology. Our completed studies in the National Science and Technology Support Program and National Key Research and Development (R&D) Program of the 12th and 13th Five-Year Plan in China found that treatment designed for specific clinical subtypes can improve the treatment effect, and meanwhile, the application of electronic-measurement based care (e-MBC) combined with smart mobile terminals can effectively provide whole-course medical management for patients, improve patient compliance and increase the efficacy of clinical diagnosis and treatment. However, due to disease diagnosis based on clinical symptomatology without subtype distinction and lack of multi-scale biological data mining, multidimensional assessment and deep integration, the results of most previous studies can hardly be used in clinical practice. Therefore, there is a strong urge to carry out a systematic research in which multidimensional evaluation of clinical characteristics and a large scale of data collection and mining are needed to form clinical diagnosis and optimal treatment regimens for depression subtypes. To achieve the goal, patients with depression will be our research subject in this study. First, on the basis of the previous cohort study and the whole-course e-MBC, patients' data of movement, respiratory rate, heart rate and sleep will be further collected. With the help of artificial intelligence (AI) technology such as deep machine learning, the data integrated with EEG imaging and specific immunometabolic markers in blood will be analyzed with clinical characteristics. The model of diagnosis and classification will be established based on multidimensional clinical assessment and verified. Second, through a prospective multicenter randomized controlled trial, optimal treatment regimens for different depression subtypes and individualized magnetic stimulation physical intervention technology navigated by AI will be explored so as to establish a predictive model of curative effect. Finally, long-term follow-up and its regular data collection can be completed on the patient diagnosis and treatment platform which is linked to the e-MBC. Thus, a stable clinical cohort and an advanced database containing multidimensional information of depression will be set up. The whole course e-MBC management platform will be optimized and promoted to improve patient compliance, treatment efficiency and prognosis. This study can provide evidence for precise diagnosis and classification of depression and optimal treatment regimens for different subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old;
2. Meeting with the criteria of major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5;
3. Scored 20 or higher on the Hamilton's Depression Scale with 24 items (HAMD-24);
4. With enough audio-visual ability and comprehensive ability to accomplish the visits;
5. No medication or washout period of at least 2 weeks
6. Scored less than 14 on the Hypomania Symptom Checklist-32 (HCL-32);

Exclusion Criteria:

1. Existing serious and active physical diseases that may interfere with treatment (abnormal indicators> 2 times the normal value), or there is a pharmacological conflict between the current medical medication and the study drug;
2. Previous mania or hypomania episodes;
3. Female patients who are pregnant, planning to be pregnant or breastfeeding;
4. Current high suicide risk (e.g. 3rd item of HAMD-24 scored≥3(suicidality));
5. Had ECT, MECT or rTMS in the past 6 months;
6. Experienced a history of dependence on psychoactive substances, organic mental disorders, personality disorders, mental retardation, neurodegenerative diseases, brain trauma and cerebrovascular diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 960 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12 weeks
  scored 7 or lower on the Hamilton's Depression Scale with 24 items

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Med-X Research Institute of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Renji Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided